CLINICAL TRIAL: NCT01229319
Title: An Investigator-Initiated Study to Assess the Safety and Efficacy of Imiquimod 3.75% Cream When Used After Cryotherapy in the Treatment of Hypertrophic Actinic Keratoses (AK) on Dorsal Hands and Forearms
Brief Title: Imiquimod 3.75% Cream in Combination With Cryotherapy in the Treatment of Hypertrophic Actinic Keratoses
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frankel, Amylynne, M.D. (Other)
Collaborators: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Gary S Goldenberg, MD/Assistant Clinical Professor Dermatology and Dermatopathology, Mount Sinai School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-0933
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis, keratocytic lesion, keratoses, cryotherapy, imiquimod
MeSH Terms: conditions — Keratosis, Actinic; Keratosis | interventions — Cryotherapy; Imiquimod

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cryo + imiquimod to Left (Experimental): Cryotherapy alone to Right arm plus cryotherapy + imiquimod 3.75% daily x 2 weeks on and 2 weeks off and 2 weeks on to Left arm
  Interventions: Drug: Cryotherapy alone to Left arm plus cryotherapy + imiquimod to Right arm
- Cryo + imiquimod to Right (Experimental): Cryotherapy alone to Left arm plus cryotherapy + imiquimod 3.75% daily x 2 weeks on and 2 weeks off and 2 weeks on to Right arm
  Interventions: Drug: Cryotherapy alone to Left arm plus cryotherapy + imiquimod to Right arm

INTERVENTIONS:
Drug: Cryotherapy alone to Left arm plus cryotherapy + imiquimod to Right arm — Cryotherapy alone to Left arm plus cryotherapy + imiquimod 3.75% daily x 2 weeks on and 2 weeks off and 2 weeks on to Right arm
  Other Names: zyclara
  Arms: cryo + imiquimod to Left
Drug: Cryotherapy alone to Left arm plus cryotherapy + imiquimod to Right arm — Cryotherapy alone to Left arm plus cryotherapy + imiquimod 3.75% daily x 2 weeks on and 2 weeks off and 2 weeks on to Right arm
  Other Names: zyclara
  Arms: Cryo + imiquimod to Right

SUMMARY:
Actinic keratoses (AK) are common cutaneous lesions associate with chronic ultraviolet radiation exposure. While most authorities consider AK as a pre-malignant lesion, some consider it as an incipient squamous cell carcinoma (SCC). In addition, the skin around clinically obvious AK lesions has been subject to the same chronic ultraviolet exposure, resulting in genetic damage and mutations, resulting in "field cancerization." Subclinical AKs may progress to clinical AKs, or even de novo invasive SCCs.

Among the current therapies for the treatment of AK are excisional surgery, cryosurgery, electrodessication and curettage, topical chemotherapy and light therapies. With cryotherapy, treated lesion clearance rates at 3 months post-treatment after double-freeze thaw cryotherapy has been reported to be around 76-88%; Overall lesion clearance rate at approximately 5 months post-cryosurgery has been reported to be 35-51%.

Imiquimod is a topical immune response modifier and a 5% formulation has been approved for the treatment of AKs in the US as a 2x/week for 16 week regimen and in Europe as a 3x/week for 4 week regimen for 1 or 2 courses of therapy. Topical imiquimod treatment may also reduce subclinical lesions in the treatment area, resulting in fewer "new" AK lesions developing over the same period of time when compared to focal treatment. In a comparison of cryosurgery versus imiquimod for the treatment of AKs, Krawtchenko et al reported initial complete clearance rates of 68 and 85% by clinical assessment, respectively. However, the treatment field sustained clearance rate was 4% versus 73%, respectively. Tan et al reported that while application of imiquimod or vehicle following cryosurgery resulted in comparable target AK clearance rates at 12 weeks of 79% versus 76%, respectively, the imiquimod group had fewer total AKs and fewer subclinical AKs.

Imiquimod cream at a concentration of 3.75% has been found in Phase 3 studies to be superior to placebo cream with respect to clearance of AKs using a regimen of up to 2 packets (250 mg of cream per packet, 500 mg total) applied daily to the entire face (approximately 200 cm2) for two 2-week treatment cycles separated by a 2-week no-treatment period. This study aims to examine the benefit of cryotherapy in combination with imiquimod 3.75% compared to cryotherapy alone.

DETAILED DESCRIPTION:
Actinic keratoses (AK) are common cutaneous lesions associate with chronic ultraviolet radiation exposure. Ultraviolet radiation produces local and systemic immunosuppression, mutations in the p53 tumor suppressor gene, and deoxyribonucleic acid pyrimidine covalent dimmers, each of which is believed to contribute to the dysplasia seen in AK. While most authorities consider AK as a pre-malignant lesion, some consider it as an incipient squamous cell carcinoma (SCC). The risk for progression to SCC for an individual AK is reportedly low but highly variable; however, as patients often have multplie AKs, the overall risk for progression over a lifetime can be significant; thus treatment of AKs is warranted. In addition, the skin around clinically obvious AK lesions has been subject to the same chronic ultraviolet exposure, resulting in genetic damage and mutations, resulting in "field cancerization." Subclinical AKs may progress to clinical AKs, or even de novo invasive SCCs.

Among the current therapies for the treatment of AK are excisional surgery, cryosurgery, electrodessication and curettage, topical chemotherapy and light therapies. With provider-administered devices, temperature utilized, times of contact, and other variations in administration, influence efficacy of treatment. Efficacy can be improved by increasing the freeze time, but this is often associated with greater discomfort, more severe skin necrosis, and increased risk of post-treatment hypopigmentation. In addition, as with other lesion-directed therapies, cryosurgery does not treat subclinical lesions in the surrounding skin. Treated lesion clearance rates at 3 months post-treatment after double-freeze thaw cryotherapy has been reported to be around 76-88%; however, new lesions in the treatment field were not included. Overall lesion clearance rate, including new subclinical lesions, at approximately 5 months post-cryosurgery has been reported to be 35-51%. There is limited information on long-term AK clearance rates after cryosurgery and those reports differ in their methods of calculation. In a study comparing cyrotherapy, imiquimod and 5-fluorouracil, at 12 months post cryotherapy 28% (7/25) had complete clearance of baseline lesions that had undergone cryotherapy, but only 4% (1/25) had complete clearance of the treatment field.

Imiquimod is a topical immune response modifier that activates the innate immune system via Toll-like receptor 7, as well as enhances the acquired immune system. A 5% topical formulation has been approved for the treatment of AKs in the US as a 2x/week for 16 week regimen and in Europe as a 3x/week for 4 week regimen for 1 or 2 courses of therapy. Topical imiquimod treatment may also reduce subclinical lesions in the treatment area, resulting in fewer "new" AK lesions developing over the same period of time when compared to focal treatment. In a comparison of cryosurgery versus imiquimod for the treatment of AKs, Krawtchenko et al reported initial complete clearance rates of 68 and 85% by clinical assessment, respectively. However, the treatment field sustained clearance rate was 4% versus 73%, respectively. Tan et al reported that while application of imiquimod or vehicle following cryosurgery resulted in comparable target AK clearance rates at 12 weeks of 79% versus 76%, respectively, the imiquimod group had fewer total AKs and fewer subclinical AKs.

The imiquimod 5% formulation has limitations for the treatment of AKs. It is approved for the treatment of a small area of skin (25 cm2), uses a less than intuitive 2 times per week (2x/week) dosing schedule, and has a prolonged treatment period (16 weeks). Dosing more frequently than 3x/week with imiquimod 5% cream was not well tolerated in subjects with AK. Imiquimod cream at a concentration of 3.75% has been found in Phase 3 studies to be superior to placebo cream with respect to clearance of AKs using a regimen of up to 2 packets (250 mg of cream per packet, 500 mg total) applied daily to the entire face (approximately 200 cm2) for two 2-week treatment cycles separated by a 2-week no-treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years old.
2. Subjects must be in good general health as confirmed by the medical history.
3. Subjects must be able to read, sign, and understand the informed consent
4. Prior to cryosurgery, subjects have at least 3 hypertrophic actinic keratoses on each dorsal hand/forearm.
5. Subject must be willing to forego any other treatments on the dorsum of the hands and or/forearms, including tanning bed use and excessive sun exposure while in the study.
6. Subject is willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up periods and to comply with all study requirements including concomitant medication and other treatment restrictions.
7. If subject is a female of childbearing potential she must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.

Exclusion Criteria:

1. Subjects with a history of melanoma anywhere on the body.
2. Subjects with an unstable medical condition as deemed by the clinical investigator.
3. Subjects with non-melanoma skin cancer on the dorsum of the hands or forearms.
4. Subjects with any dermatologic disease in the treatment area that may be exacerbated by the treatment proposed or that might impair the evaluation of AKs.
5. Subjects who have previously been treated with imiquimod: on the dorsum of the hands or forearms in the past 6 months; or outside of the study area within the past 30 days.
6. Women who are pregnant, lactating, or planning to become pregnant during the study period.
7. Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc).
8. Subjects who have active chemical dependency or alcoholism as assessed by the investigator.
9. Subjects who have known allergies to any excipient in the study cream.
10. Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device on the study area within 30 days prior to study treatment initiation.
11. Subjects who have received any of the following within 90 days prior to study treatment initiation:

    * interferon or interferon inducers
    * cytotoxic drugs
    * immunomodulators or immunosuppressive therapies (inhaled/ intranasal steroids are permitted)
    * oral or parenteral corticosteroids
    * topical corticosteroids if greater than 2 gm/day
    * any dermatologic procedures or surgeries on the study area (including any AK treatments)
12. Subjects who have used any topical prescription medications on the study area within 30 days prior to study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Clearance of Actinic Keratoses | 14 weeks
  AK lesion count, photography

SECONDARY OUTCOMES:
Local Skin Reactions (LSRs) | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Goldenberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, Department of Dermatology, Clinical Trials, New York, New York, United States